CLINICAL TRIAL: NCT03908658
Title: The Effectiveness of Inspiratory Muscle Training and Nasal High Flow Oxygen in Difficult Weaning of ICU Patients
Brief Title: Inspiratory Muscle Training and Nasal High Flow in Difficult Weaning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, ISCHAKI ELENI, Consultant, ICU Department, Evangelismos Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6345/14-03-2019
Record Dates: First submitted 2019-04-04; First posted 2019-04-09 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: High-risk for Reintubation Patients; Weaning Outcome
Keywords: inspiratory muscle training; Nasal High Flow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training and Nasal High Flow (Active Comparator): Inspiratory Muscle Training will start as soon as the patient wakes up and is cooperative, ventilated with support settings. Nasal High Flow will be applied immediately after extubation. IMT intervention will continue until patient's discharge from the ICU
  Interventions: Other: Inspiratory muscle Training and Nasal High Flow
- Inspiratory Muscle Training and Venturi mask (Active Comparator): IMT will start as soon as the patient wakes up and is cooperative, ventilated with support settings. Venturi mask will be applied immediately after extubation. IMT intervention will continue until patient's discharge from the ICU
  Interventions: Device: Inspiratory muscle training and Venturi mask

INTERVENTIONS:
Other: Inspiratory muscle Training and Nasal High Flow — Inspiratory muscle Training will be used to increase respiratory muscle strength. Initial settings will depend on patient's maximal inspiratory pressure. Nasal High Flow will support respiratory muscles and thus reduce the work of breathing. By this mechanism the endurance of the respiratory muscles will increase in parallel with the strenght
  Arms: Inspiratory Muscle Training and Nasal High Flow
Device: Inspiratory muscle training and Venturi mask — Inspiratory muscle Training will be used to increase respiratory muscle strength. Initial settings will depend on patient's maximal inspiratory pressure. Venturi mask is usually applied after extubation in every day clinical practice for oxygen supplementation
  Arms: Inspiratory Muscle Training and Venturi mask

SUMMARY:
The purpose of the present study is to investigate the effectiveness of inspiratory muscle training and nasal high flow oxygen in patients with difficult weaning and high-risk for re-intubation. The hypothesis of the study is that starting inspiratory muscle training once patients are awake and co-operative along with the application of nasal high flow oxygen immediately after extubation will have a beneficial effect in preventive re-intubation in these high-risk patients.

DETAILED DESCRIPTION:
20-30% of intubated patients are difficult to be weaned off the mechanical ventilation and have a prolonged ICU stay. It is well established that prolonged ICU stay is associated with reduced muscle strength, functional ability and quality of life.

Inspiratory muscle training (IMT) via a threshold device has been proposed as an effective exercise for minimizing the detrimental effect of mechanical ventilation in critical ill patients with prolonged weaning. Additionally, Nasal High Flow (NHF) oxygen has been proved to support efficiently either high or low-risk patients after extubation and thus preventing re-intubation.

A randomized intervention study was designed to assess the efficacy of combining IMT and NHF as therapeutic strategies for difficult weaning. Once patients with prognostic factors of difficult weaning are awake and co-operative they will be randomized to one of the two following study groups: 1) IMT and NHF group, 2) IMT and Venturi mask group. IMT will start as soon as the patient wakes up and is cooperative, ventilated with support settings. Each allocated oxygen delivery device will be applied immediately after extubation. IMT intervention will continue until patients' discharge from the ICU.

ELIGIBILITY:
Inclusion Criteria:

* >65 years,
* BMI> 35kg/m2,
* weak cough,
* heart (i.e heart failure ) and lung comorbidities (i.e COPD),
* hypercapnia during mechanical ventilation
* > 72hours on mechanical ventilation
* failed first spontaneous breathing trial

Exclusion Criteria:

* Glasgow Coma scale (GCS)<13,
* pre-existing neuromuscular disease or deformity of Spinal Cord,
* terminal disease
* hemodynamic instability with >0.1μg/kg/min noradrenaline
* patients of immediately need of Non-invasive ventilation after extubation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-03-20 (Estimated)

PRIMARY OUTCOMES:
Rate of weaning failure | 48 hours after extubation
  Rate of weaning failure in high-risk for reintubation patients

SECONDARY OUTCOMES:
Maximal Inspiratory Pressure | Within 2 hours after patient randomization, within 24 hours after extubation, within 24 hours after ICU discharge
  Maximal Inspiratory Pressure (MIP) will be assessed witn an unidirectional expiratory valve which permit exhalation while inspiration is blocked. One side of the valve will be attached to the patient's endotracheal tube and the other side to a manometer. Manometer could register pressures from 0 to 60 cmH20. Patients will be disconnected from the ventilator and attached to the valve for a period of more than 30 sec. The most negative value will be recorded
Maximal Expiratory Pressure | Within 2 hours after patient randomization, within 24 hours after extubation, within 24 hours after ICU discharge
  Maximal Expiratory Pressure (MEP) will be assessed witn an unidirectional inspiratory valve which permit inspiration while expiration is blocked. One side of the valve will be attached to the patient's endotracheal tube and the other side to a manometer. Manometer could register pressures from 0 to 60 cmH20. Patients will be disconnected from the ventilator and attached to the valve for a period of more than 30 sec. The highest value will be recorded
Endurance of respiratory muscles | Within 2 hours after patient randomization, within 24 hours after extubation , within 24 hours after ICU discharge
  Endurance of respiratory muscles will be calculated comparing the preloading and postloading values of the MIP
Muscle strenght | Within 2 hours after patient randomization, within 24 hours after ICU discharge, within 24 hours before hospital discharge
  Muscle strength will be assessed by the sum of Medical Research Council (MRC) scale for muscle strength in 6 different muscle groups ( shoulder abductors, forearm flexors, wrist flexors, hip flexors, knee extensors and plantar dorsiflexors) for both body sides. Each muscle group scores from 0 (no contraction) up to 5 (movement against gravity) and the total score range from 0 (worse outcome) up to 60 (best outcome)
Functional ability | Within 24 hours after ICU discharge, within 24 hours before hospital discharge
  Functional ability will be assessed by Functional Independence Measure (FIM) which includes 18 questions (13 motor tasks and 5 cognitive tasks). Each item is scored on a 7 point ordinal scale, ranging from a score of 1 (total inability-dependence) to a score of 7 (total independence). The higher the score, the more independent the patient is in performing the task associated with that item.The total score for the FIM motor subscale (the sum of the individual motor subscale items) will be a value between 13 and 91. The total score for the FIM cognition subscale (the sum of the individual cognition subscale items) will be a value between 5 and 35. The total score for the FIM instrument (the sum of the motor and cognition subscale scores) will be a value between 18 (total dependency) and 126 total indepedency
Short Form 36 Health Survey (SF-36) questionnaire | Within 24 hours before hospital discharge
  Quality of life (QoL) will be assessed by Short Form 36 Health Survey (SF-36) which includes 36 items to measure 8 QoL domains. More specifically, from SF-36 only the domains parts of Physical Functioning (PF) which includes 10 questions with possible scores from 1 to 3, the Role Physical (RF) which includes 4 yes or no questions, the Social Functioning (SF) which includes 2 questions with possible scores form 1 to 5 and the Mental Health domain (MH) which includes 9 questions with possible scores form 1 to 9 will be used. Regarding the scoring of the questions 1 is the worst outcome. Each domain is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Euro-Qol 5 Dimensions 5 Level of severity scale (Euro-Qol 5D-5L scale) | Within 24 hours before hospital discharge
  Euro-Qol 5D-5L questionnaire includes 5 domains and an optic analogue scale from 0 (worse) up to 100 (best). Each domain (mobility, self care, usual activities, pain / discomfort, anxiety / depression) scores from 1(best score) up to 5 (worse score). The total score of all domains ranges from 5 (best score) up to 25 (worse score).The total perceived quality of life will be graded by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelismos Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
Participants' data will be available will be available following publication
Supporting Information: Study Protocol, CSR
Time Frame: following publication